CLINICAL TRIAL: NCT06306612
Title: Systemic Therapy Combined With Cytoreductive Prostatectomy for the Treatment of de Novo Poly-metastatic Hormone Sensitive Prostate Cancer: A Prospective, Open-label Randomized Controlled Trial
Brief Title: CytoREductive prostAtectomy for Poly-metastatic Hormone sensiTIVE Prostate Cancer
Acronym: CREATIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Liang Dong, Associate Research Fellow, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-0165
Record Dates: First submitted 2024-02-19; First posted 2024-03-12 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group start with 6 cycles of induction chemohormonal therapy followed with cytoreductive prostatectomy and postoperative adjuvant radiotherapy if needed. All patients continued maintenance therapy.
  Interventions: Drug: Systemic Chemohormonal Therapy; Drug: Systemic Hormonal Therapy; Procedure: Cytoreductive Prostatectomy; Procedure: Postoperative Adjuvant Radiotherapy
- Control group (Active Comparator): The control group start with 6 cycles of chemohormonal therapy followed by continued maintenance therapy.
  Interventions: Drug: Systemic Chemohormonal Therapy; Drug: Systemic Hormonal Therapy

INTERVENTIONS:
Drug: Systemic Chemohormonal Therapy — Under continuous ADT, docetaxel 75mg/m^2 body surface area every 21 days, oral dexamethasone 7.5mg pretreatment 12h, 3h, 1h before each infusion of docetaxel, and a total of 10mg of prednisolone per day when needed according to the decision of the researcher (in the case of grade 3 and above neutropenia or peripheral edema); oral darolutamide 600mg twice per day, 21 days for one cycle, six cycles in total.
Drug: Systemic Hormonal Therapy — Under continuous ADT, oral darolutamide 600mg twice per day
Procedure: Cytoreductive Prostatectomy — Cytoreductive prostatectomy was performed after six cycles of neoadjuvant systemic chemohormonal therapy.
  Arms: Experimental group
Procedure: Postoperative Adjuvant Radiotherapy — Postoperative adjuvant radiotherapy of prostate bed is performed, if margin positive, with conventional segmentation and the dose of 64-72Gy.
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to compare systemic therapy combined with cytoreductive prostatectomy with standard of care (SOC) in de novo poly-metastatic hormone sensitive prostate cancer (de novo pmHSPC). The main questions it aims to answer are:

1. To explore the clinical benefit and safety of systemic therapy combined with cytoreductive prostatectomy for patients with de novo pmHSPC.
2. To explore the characteristics of the subgroup of patients who could benefit more from the above treatment.
3. To explore the relationship between stage efficacy and clinical prognosis.
4. To explore the correlation between molecular imaging such as PSMA-PET/CT and its changes with treatment efficacy.

Participants will undergo systemic therapy combined with cytoreductive prostatectomy.

Researchers will compare systemic therapy combined with cytoreductive prostatectomy with SOC to see the pros and cons of the two strategies.

DETAILED DESCRIPTION:
1. Subject Management

1. Recruitment of subjects The subjects are recruited from the outpatient clinic of the Department of Urology of Renji Hospital, Shanghai Jiao Tong University School of Medicine; the specific time was from the beginning of the recruitment of subjects to the end of reaching the target of the recruitment of subjects. If the attending physician's initial judgment meets the criteria for NAC, recruitment will be carried out after communicating with the patient and his/her family.
2. Informed consent process After the attending physician (investigator) finds patients who initially meet the enrollment criteria of this trial, he/she should give a written and verbal explanation to the subjects about the background, nature, significance, steps, benefits, risks, compensation, injury compensation, and withdrawal of the study, and he/she must obtain an informed consent form signed by each subject (or subject's legal representative). The informed consent form is dated, and the informed consent form and its copy are kept separately by the investigator and the subject.
3. Checking the enrollment criteria As soon as possible after the preliminary identification of subjects, the attending physician and the investigator will check the enrollment criteria together, make a formal decision to recruit or not to recruit into the group and inform the subjects, and explain the reasons for not recruiting into the group in detail and record them.
4. Examination of medical history and records of combined medications During the initial screening and verification of the enrollment criteria, the attending physician will obtain the subject's past history, current medical history, personal history, as well as comorbid medications, and previous medications. If necessary, the history and co-medication records will be declared by the patient himself/herself or under the supervision of the attending physician while signing the informed consent form.
5. Assignment of screening number At the time of signing the informed consent, each patient is assigned a screening number, the rules for the preparation of the screening number are specified separately, and should ensure the principles of continuity, traceability and de-specialization.
6. Assignment of treatment/randomization group numbers Sequence generation: the data manager should use SAS statistical software (SAS Institute. Cary, NC, USA) to generate the allocation sequence in a stratified block randomization with block length set to 4. All subjects were randomly (1:1) assigned to trial and control groups. Factors for stratification included tumor stage (M1a/M1b/M1c) and baseline alkaline phosphatase level (greater/less than ULN). Randomized assignment sequences were performed using sequentially coded sequestration, and interventions should in principle be assigned as soon as possible after generation of the randomized assignment sequence. Sequences should not be accessed by anyone other than the restricted data manager prior to allocation of the intervention.

   Implementation: Generation of the randomized allocation sequence and allocation of the intervention by the data manager, and the generation of the sequence and the allocation of the intervention should be performed by different managers; recruitment of subjects by the attending clinical physician (investigator).
7. Trial Adherence Management During the course of the trial, patients' adherence to the trial will be examined and documented by the supervising physician at each visit and as deemed necessary by the investigator. If necessary, subjects may be instructed to complete a medication diary, which will be checked by the supervising physician and the investigator at each visit. Adherence reports are submitted to the Ombudsman for review as deemed necessary.

2. Intervention Trial group: Systemic therapy plus cytoreductive prostatectomy Control group: Standard of care.

3. Efficacy measurement Efficacy measurements of the specified items and frequencies are performed according to the visit requirements, and the efficacy is observed and recognized strictly according to the criteria set out in the outcomes, and the investigators and evaluators should form an efficacy report and include it in the case report form. PET-CT and PSMA-PET/CT examinations were for the exploratory purpose of this study, so they could be performed on a voluntary basis at the subjects' own expense and with their fully informed consent. The performance or failure of the examination and its results should not affect the performance of other treatments, nor should it affect the performance of other visits and programs.

In order to ensure the objectivity and comparability of the assessment of outcome indicators, the grouping information was hidden from the imaging evaluators and laboratory technicians, and for the scale-based visits, the patient self-assessment was used as the primary method, supplemented by the evaluation under the guidance of the professional staff, and the grouping information was hidden from the supervisory staff when the latter method was used.

4. Data Management

1. Data entry The investigator loads the data into the case report form in a timely, complete, correct and legible manner based on the subject's original observation record. The questionnaire after review and signature by the supervisor should be sent to the Clinical Research Data Manager in a timely manner. The entry is done using the appropriate database system of two-person dual-machine entry, after which the database is compared twice, during which if any problems are found, the supervisor is promptly notified and the researcher is asked to make an answer. The exchange of all kinds of questions and answers between them should be in the form of a questionnaire, which should be kept for reference.
2. Content and manner of data verification and management When all the case report forms have been double-entered and checked for accuracy, a database check report will be written by the data manager, which will include study completion (including list of dislodged subjects), inclusion/exclusion criteria check, completeness check, logical consistency check, outlier data check, time-window check, combined medication check, and adverse event check. At the audit meeting, the principal investigator, representatives of the sponsor, supervisors, data managers and statisticians will make a resolution on the issues raised in the subjects' signing of the informed consent form and the database checking report, write an audit report, and the database will be locked at the same time.
3. Data archiving The case report form, after data entry and verification are completed as required, will be filed and stored in numbered order and filled with search catalogs, etc., for examination. Electronic data files including databases, examination procedures, analytical procedures, analytical results, codebooks and description documents should be classified and kept with multiple backups on different disks or recording media for proper preservation and prevention of damage. All original files should be kept for the period within the corresponding regulations.

5. Analysis and statistical methods Before the start and after the end of each phase of the trial and the trial, the principal investigator, representatives of the sponsor, supervisors, data administrators and statisticians should carry out internal data analysis, including the completion of the study (including the list of dislodged subjects), analysis of the efficacy of the phase, and analysis of the adverse events, etc., and submit the analysis report to the review meeting for consideration.

According to the basic principle of Intention-to-Treat (ITT), the analysis of the main indicators should include all randomized subjects, regardless of whether they completed the trial or not. Therefore, this study used the full analysis set for analysis; when choosing the full analysis set for statistical analysis, the missing of the main indicators should be avoided as much as possible, and when the indicators are indeed missing, the deletion and the reason for deletion should be indicated in the analysis, and the mixed-effects model of repeated-measures data should be applied in the statistical analysis for processing.

Statistical analyses included stage efficacy analyses and summative efficacy analyses. Stage analysis was conducted after all subjects had completed the induction/chemotherapy phase and after all subjects in the trial group had completed the topical treatment phase. Terminal statistical analysis was conducted after all subjects had reached the primary endpoint of the study or had completed 3 years or had been discontinued/withdrawn, i.e., had completed the maintenance phase, and the trial had been completed. Statistical analyses were conducted to determine the relationship between subjects' achievement of the primary and secondary trial endpoints at each stage, and the stage-specific changes in each of the visits associated with the trial endpoints, and their potential impact on factors including, but not limited to, baseline status, receipt of the intervention, and changes in other visits. Statistical analyses were performed according to the following specifications:

Statistical descriptions of patients' baseline clinical characteristics; hypothesis testing for outcomes that manifested as categorical variables and those that manifested as ordered categorical variables using chi-square, Fisher's exact test, and rank-sum tests, as necessary; analysis of outcome indicators of a survival nature using Kaplan-Meier survival analysis; and exploration of the influence of each potentially influencing factor on the outcome using univariate and multivariate Cox regression. The impact of potential influences on outcomes was explored using univariate and multivariate Cox regression.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose of this trial and sign a written informed consent;
2. Men aged 18-85 years;
3. have histologically or cytologically confirmed adenocarcinoma of the prostate;
4. Have multiple metastatic disease, defined as follows: according to RECIST v1.1, metastatic disease was defined as metastatic foci detected on bone scans or measurable lymph nodes or soft tissue or visceral lesions above the aortic bifurcation. Lymph nodes were defined as measurable if their short-axis diameter was ≥15 mm; soft tissue/visceral lesions were defined as measurable if their long-axis diameter was ≥10 mm. and total number of metastatic lesions ≥ 5. Patients with only regional lymph node metastases (N1, below the aortic bifurcation) were not eligible for the study.
5. At the investigator's discretion, patients must meet the indications for ADT and docetaxel;
6. Patients have not received any prior local or systemic therapy for prostate cancer primary or metastasis.
7. Eastern Cooperative Oncology Group (ECOG) score of 0-1;
8. Blood count at screening: hemoglobin ≥ 9.0 g/dL, absolute neutrophil count ≥ 1.5 x 10^9/L, and platelet count ≥ 100 x 10^9/L (patient has not received any colony-stimulating factor within 4 weeks or a transfusion or blood product within 7 days prior to blood collection)
9. Serum alanine aminotransferase and/or aspartate aminotransferase ≤ 1.5 x Upper limit of normal (ULN), total bilirubin ≤ ULN, creatinine ≤ 2.0 x ULN.

Exclusion Criteria:

1. Prior therapy: ADT, second-generation androgen receptor inhibitors, CYP17 enzyme inhibitors, any chemotherapy or immunotherapy for prostate cancer, radiotherapy (external radiation radiotherapy, brachytherapy, or radiopharmaceuticals);
2. Known hypersensitivity to any of the investigational drugs, or excipients in the preparations;
3. Contraindication to CT/MRI examination;
4. Any of the following conditions within 6 months prior to randomization: stroke, myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass grafting, or congestive heart failure (New York Heart Association cardiac function class III or IV);
5. uncontrolled hypertension as evidenced by a resting systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 100 mm Hg after treatment
6. History of prior malignancy, except basal cell or cutaneous squamous cell carcinoma in complete remission;
7. History of gastrointestinal disorders or surgery expected to significantly interfere with the absorption of study drug(s);
8. Active acute and chronic viral hepatitis, known HIV infection;
9. Prior (28 days prior to initiation of study drug or 5 half-lives of investigational therapy from a prior study, whichever is longer) or concurrent participation in another clinical study of study drug;
10. Any other serious or unstable medical condition or condition that may interfere with their participation in the study or the evaluation of study results or may jeopardize the safety of the trial and other conditions;
11. Inability to swallow oral medications;
12. A close interest in the research center.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Castration resistant-free survival | Through study completion, assessed up to three years.
  From date of randomization to the date of the following events, whichever occurs first: prostate specific antigen (PSA) elevation above nadir of at least 2 ng/mL or elevation above nadir of at least 25% when testosterone is at castration level (<50 ng/dL), as determined by reassessment at least 3 weeks later; or soft tissue, visceral, or radiographic progression of skeletal lesions: as recommended by the Prostate Cancer Clinical Trials Working Group (PCWG)3, Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 is applied via magnetic resonance imaging (MRI) of the thorax/abdomen/pelvis to determine radiographic progression of soft tissue/visceral lesions; bone metastases are identified separately from soft tissue/visceral metastases and are determined by 99mTc methylenediphosphonate bone scanning of the whole body according to PCWG3. Metastases may also be identified using PSMA-PET/CT.

SECONDARY OUTCOMES:
Overall Survival | Through study completion, assessed up to three years.
  From date of randomization until the date of death from any cause.
PSA response | Through study completion, assessed up to three years.
  Complete remission is defined as PSA detectable (≥0.2 ng/mL) at baseline and undetectable (<0.2 ng/mL) for the duration of the study; PSA50, and PSA90 response are defined as a ≥50% or ≥90% decrease in the measured PSA level from baseline to post-baseline as determined by reassessment after at least 3 weeks.
Symptomatic skeletal event | Through study completion, assessed up to three years.
  Defined as external radiation therapy for the relief of skeletal symptoms, a new symptomatic pathologic fracture or vertebral compression fracture or related orthopedic surgical intervention, or death, whichever occurred first.
Pain progression | Through study completion, assessed up to three years.
  Pain is assessed at each visit using the Visual Analogue Scale (VAS). Pain progression is defined as an increase of ≥2 points from the nadir of the worst pain score or opioid use for more than 7 consecutive days in two consecutive assessments ≥4 weeks apart for asymptomatic patients ("worst pain in 24 hours" score of 0 at baseline). For symptomatic patients (worst pain in 24 hours" score >0 at baseline), pain progression was defined as an increase of ≥2 points from the nadir of the worst pain score on two consecutive assessments ≥4 weeks apart and with a worst pain score of ≥4 or or initiation of short-acting or long-acting opioid therapy for cancer pain for more than 7 consecutive days.
Deterioration of disease-related somatic symptoms | Through study completion, assessed up to three years.
  According to the National Comprehensive Cancer Network/Functional Assessment of Cancer Care Prostate Cancer Symptom Index 17-item questionnaire (NCCN-FACT FPSI-17), worsening of disease-related somatic symptoms was defined as a 3-point decrease in the Disease-related Somatic Symptoms subscale (FPSI-DRS-P subscale) from baseline on two consecutive assessments ≥4 weeks apart.

OTHER OUTCOMES:
Pathological and molecular response | At baseline and at the end of the 6th cycle of induction chemohormonal therapy (each cycle is 21 days).
  Tissue samples are collected and closely examined by pathologists to assess patients' baseline pathological stage as well as their pathological response after induction systemic therapy. Also, tissue samples and paired body fluid samples are retained under appropriate conditions for future exploratory studies (including but not limited to transcriptomics, proteomics, metabolomics sequencing on single-cell and bulk level, SRT and EV-related studies) concerning molecular characteristics and response to therapy. Informed consent form is required prior to collection of above-mentioned samples.

CONTACTS AND LOCATIONS:
Overall Officials: Yinjie Zhu, Dr., Principal Investigator — RenJi Hospital; Liang Dong, Dr., Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Background] Mohler JL, Antonarakis ES, Armstrong AJ, D'Amico AV, Davis BJ, Dorff T, Eastham JA, Enke CA, Farrington TA, Higano CS, Horwitz EM, Hurwitz M, Ippolito JE, Kane CJ, Kuettel MR, Lang JM, McKenney J, Netto G, Penson DF, Plimack ER, Pow-Sang JM, Pugh TJ, Richey S, Roach M, Rosenfeld S, Schaeffer E, Shabsigh A, Small EJ, Spratt DE, Srinivas S, Tward J, Shead DA, Freedman-Cass DA. Prostate Cancer, Version 2.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 May 1;17(5):479-505. doi: 10.6004/jnccn.2019.0023. PMID 31085757
- [Background] Schaeffer EM, Srinivas S, Adra N, An Y, Barocas D, Bitting R, Bryce A, Chapin B, Cheng HH, D'Amico AV, Desai N, Dorff T, Eastham JA, Farrington TA, Gao X, Gupta S, Guzzo T, Ippolito JE, Kuettel MR, Lang JM, Lotan T, McKay RR, Morgan T, Netto G, Pow-Sang JM, Reiter R, Roach M, Robin T, Rosenfeld S, Shabsigh A, Spratt D, Teply BA, Tward J, Valicenti R, Wong JK, Berardi RA, Shead DA, Freedman-Cass DA. NCCN Guidelines(R) Insights: Prostate Cancer, Version 1.2023. J Natl Compr Canc Netw. 2022 Dec;20(12):1288-1298. doi: 10.6004/jnccn.2022.0063. PMID 36509074
- [Background] Ploussard G, Fossati N, Wiegel T, D'Amico A, Hofman MS, Gillessen S, Mottet N, Joniau S, Spratt DE. Management of Persistently Elevated Prostate-specific Antigen After Radical Prostatectomy: A Systematic Review of the Literature. Eur Urol Oncol. 2021 Apr;4(2):150-169. doi: 10.1016/j.euo.2021.01.001. Epub 2021 Feb 8. PMID 33574012
- [Background] Pound CR, Partin AW, Epstein JI, Walsh PC. Prostate-specific antigen after anatomic radical retropubic prostatectomy. Patterns of recurrence and cancer control. Urol Clin North Am. 1997 May;24(2):395-406. doi: 10.1016/s0094-0143(05)70386-4. PMID 9126237
- [Background] Trapasso JG, deKernion JB, Smith RB, Dorey F. The incidence and significance of detectable levels of serum prostate specific antigen after radical prostatectomy. J Urol. 1994 Nov;152(5 Pt 2):1821-5. doi: 10.1016/s0022-5347(17)32394-7. PMID 7523728
- [Background] Efstathiou E, Davis JW, Pisters L, Li W, Wen S, McMullin RP, Gormley M, Ricci D, Titus M, Hoang A, Zurita AJ, Tran N, Peng W, Kheoh T, Molina A, Troncoso P, Logothetis CJ. Clinical and Biological Characterisation of Localised High-risk Prostate Cancer: Results of a Randomised Preoperative Study of a Luteinising Hormone-releasing Hormone Agonist with or Without Abiraterone Acetate plus Prednisone. Eur Urol. 2019 Oct;76(4):418-424. doi: 10.1016/j.eururo.2019.05.010. Epub 2019 Jun 6. PMID 31176622
- [Background] Connor MJ, Shah TT, Horan G, Bevan CL, Winkler M, Ahmed HU. Cytoreductive treatment strategies for de novo metastatic prostate cancer. Nat Rev Clin Oncol. 2020 Mar;17(3):168-182. doi: 10.1038/s41571-019-0284-3. Epub 2019 Nov 11. PMID 31712648
- [Background] Powell IJ, Tangen CM, Miller GJ, Lowe BA, Haas G, Carroll PR, Osswald MB, DeVERE WHITE R, Thompson IM Jr, Crawford ED. Neoadjuvant therapy before radical prostatectomy for clinical T3/T4 carcinoma of the prostate: 5-year followup, Phase II Southwest Oncology Group Study 9109. J Urol. 2002 Nov;168(5):2016-9. doi: 10.1016/S0022-5347(05)64285-1. PMID 12394698
- [Background] Gratzke C, Engel J, Stief CG. Role of radical prostatectomy in metastatic prostate cancer: data from the Munich Cancer Registry. Eur Urol. 2014 Sep;66(3):602-3. doi: 10.1016/j.eururo.2014.04.009. Epub 2014 May 10. No abstract available. PMID 24821581
- [Background] Heidenreich A, Pfister D, Porres D. Cytoreductive radical prostatectomy in patients with prostate cancer and low volume skeletal metastases: results of a feasibility and case-control study. J Urol. 2015 Mar;193(3):832-8. doi: 10.1016/j.juro.2014.09.089. Epub 2014 Sep 22. PMID 25254935
- [Background] Buelens S, Poelaert F, Claeys T, De Bleser E, Dhondt B, Verla W, Ost P, Rappe B, De Troyer B, Verbaeys C, Kimpe B, Billiet I, Plancke H, Fransis K, Willemen P, Ameye F, Decaestecker K, Lumen N. Multicentre, prospective study on local treatment of metastatic prostate cancer (LoMP study). BJU Int. 2022 Jun;129(6):699-707. doi: 10.1111/bju.15553. Epub 2021 Aug 8. PMID 34289231
- [Background] Parker CC, James ND, Brawley CD, Clarke NW, Hoyle AP, Ali A, Ritchie AWS, Attard G, Chowdhury S, Cross W, Dearnaley DP, Gillessen S, Gilson C, Jones RJ, Langley RE, Malik ZI, Mason MD, Matheson D, Millman R, Russell JM, Thalmann GN, Amos CL, Alonzi R, Bahl A, Birtle A, Din O, Douis H, Eswar C, Gale J, Gannon MR, Jonnada S, Khaksar S, Lester JF, O'Sullivan JM, Parikh OA, Pedley ID, Pudney DM, Sheehan DJ, Srihari NN, Tran ATH, Parmar MKB, Sydes MR; Systemic Therapy for Advanced or Metastatic Prostate cancer: Evaluation of Drug Efficacy (STAMPEDE) investigators. Radiotherapy to the primary tumour for newly diagnosed, metastatic prostate cancer (STAMPEDE): a randomised controlled phase 3 trial. Lancet. 2018 Dec 1;392(10162):2353-2366. doi: 10.1016/S0140-6736(18)32486-3. Epub 2018 Oct 21. PMID 30355464
- [Background] Eastham JA, Heller G, Halabi S, Monk JP 3rd, Beltran H, Gleave M, Evans CP, Clinton SK, Szmulewitz RZ, Coleman J, Hillman DW, Watt CR, George S, Sanda MG, Hahn OM, Taplin ME, Parsons JK, Mohler JL, Small EJ, Morris MJ. Cancer and Leukemia Group B 90203 (Alliance): Radical Prostatectomy With or Without Neoadjuvant Chemohormonal Therapy in Localized, High-Risk Prostate Cancer. J Clin Oncol. 2020 Sep 10;38(26):3042-3050. doi: 10.1200/JCO.20.00315. Epub 2020 Jul 24. PMID 32706639
- [Background] Smith MR, Hussain M, Saad F, Fizazi K, Sternberg CN, Crawford ED, Kopyltsov E, Park CH, Alekseev B, Montesa-Pino A, Ye D, Parnis F, Cruz F, Tammela TLJ, Suzuki H, Utriainen T, Fu C, Uemura M, Mendez-Vidal MJ, Maughan BL, Joensuu H, Thiele S, Li R, Kuss I, Tombal B; ARASENS Trial Investigators. Darolutamide and Survival in Metastatic, Hormone-Sensitive Prostate Cancer. N Engl J Med. 2022 Mar 24;386(12):1132-1142. doi: 10.1056/NEJMoa2119115. Epub 2022 Feb 17. PMID 35179323
- [Background] 中国医促会泌尿健康促进分会, 中国研究型医院学会泌尿外科学专业委员会. 腹腔镜(含机器人辅助)前列腺癌根治术安全共识. 现代泌尿外科杂志. 2020;25(7):575-84.
- [Background] 中国医疗保健国际交流促进会泌尿健康促进分会, 中国研究型医院学会泌尿外科学专业委员会. 前列腺癌新辅助治疗安全共识. 现代泌尿外科杂志. 2023;28(1):18-23,8.
- [Background] 中华医学会泌尿外科学分会, 中国前列腺癌联盟. 转移性前列腺癌化疗中国专家共识(2019版). 中华泌尿外科杂志. 2019;40(10):721-5.
- [Background] 中国医促会泌尿健康促进分会, 中国研究型医院学会泌尿外科学专业委员会. 前列腺癌放射治疗安全共识. 现代泌尿外科杂志. 2019;24(5):336-46.